CLINICAL TRIAL: NCT04059315
Title: Epidemiology of Oral and Maxillofacial Trauma in Province 2, Nepal
Acronym: PI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Dr Saroj Prasad Deo, Associate Professor and HOD of oral and maxillofacial surgery, Tribhuvan University, Nepal
Other Study IDs: 397-2019
Record Dates: First submitted 2019-07-31; First posted 2019-08-16 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Oral and Maxillofacial Injuries
Keywords: motor vehicle accident, epidemiology, facial fracture
MeSH Terms: conditions — Maxillofacial Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cross sectional study: This is an Epidemiological observational analytic study where the subjects sustained with oral and maxillofacial trauma will be divided into the two-time-frame;
  1st, retrospective study between 1 June 2011 to 31 May 2019
  Interventions: Other: surgical treatment of facial bone fracture
- Prospective cohort study: 2nd prospective study on 1 June 2019 to 1 June 2021.
  Interventions: Other: surgical treatment of facial bone fracture

INTERVENTIONS:
Other: surgical treatment of facial bone fracture — oral and maxillofacial injury patients admitted in our hospital. patients are getting treatment of soft and bone frature as follow soft tissue repaire, IMF, ORIF, consrvative.

SUMMARY:
Trauma is one of the leading causes of death among people under 40 years of age, the causes are numerous but the majorities are involved in road traffic accidents (RTA). The oral and maxillofacial injuries are the common presentation of hospitals either as an isolated injury ( 50%) and rest 20-30% are associated with multiple injuries to the head, neck, chest, abdomen and extremities. These injuries may cause serious functional, psychological, physical, and cosmetic disabilities.

Maxillofacial fractures are a large public health problem with a significant negative impact on an individual's overall health and even survival. The cause, severity, and temporal distribution of maxillofacial trauma can assist in establishing clinical and research priorities for effective treatment and prevention of these injuries. Also understanding maxillofacial trauma helps to evaluate the behaviour patterns of people in different countries and to establish effective prevention and treatment strategies.

To this end, numerous studies have been carried out to explore the epidemiological features of maxillofacial fractures in different population groups. However, to best our knowledge, there is a lack of research about maxillofacial injuries for this region. Hence the main purpose of this study is to investigate the epidemiological characteristics of prevalence, aetiology, sex and age distributions, fracture site, treatment pattern, associated injuries, and complications of maxillofacial fractures treated at the National Medical College and others Hospitals of Birgunj Metropolitan city over a 10-year period from June 2011 to June 2021. A specific form (oral and maxillofacial injury proforma) will be used to collect the data from medical records of patients who had sustained oral and maxillofacial injuries and admitted as well managed at the hospitals (National Medical College and Teaching Hospital, Birganj health care, Gandak hospital, LS Neuro hospital. Birgunj). Subjects would be the patients' data's/ medical records present in hospitals, Birganj. From the patient files or medical records, following information will be gathered include demographics (e.g. age, sex), the aetiology of injury, anatomic site of the fracture, time of hospital admission and operation, presence and location of associated injuries, treatment pattern, length of in-hospital stay, and complications.

DETAILED DESCRIPTION:
Introduction:

Trauma-related injuries claimed approximately 5 million lives in the world in 2016; is one of the leading causes of death among people in different age groups depending upon the causes of injuries (WHO, 2018a). More than quarters (29%) of these deaths were due to a road traffic accident. Low-income countries had the highest mortality rate due to a road traffic accident with 29.4 deaths per 100 000 population (WHO, 2018b). Many factors affect mortality rate and outcome after trauma (Kieser J et al 2002; Johnson J etal. 2012). Nature and severity of the injuries on the body part are the main factors for mortality of injured person. Among the mortality; fatality rate is 50 % within a few minutes of trauma due to damage to the brain or spinal cord or heart or major vessel or organ. Another factor affecting mortality is the standard of surgical care in the hospital; 30% die in the hospital a few hour injuries due to hypoxia and haemorrhage (hypovolemic shock). Late mortality is seen within a day to a week in hospital (20%) due to sepsis and multiorgan failure (Kovacs G, Sowers N., 2018; Prathigudupu RS et al.,2018; ).

Oral and Maxillofacial trauma is a common presentation in Emergency departments (ED) of the hospitals (Kieser J et al 2002; Wong NH etal 2012; Calderoni DR etal 2011; Katarzyna B etal 2010). Age of the patient, concomitant head injuries, airway obstruction, a pattern of facial bone fracture and increased bleeding are some of the variables of increasing death rates after maxillofacial trauma (Katarzyna B etal 2010; Kovacs G, Sowers N., 2018). Multiple body part injuries are often associated with oral and maxillofacial injuries in severely injured trauma patients(Kieser J et al, 2002; Wong NH etal, 2012; Calderoni DR etal, 2011; Katarzyna B etal. 2010; Prathigudupu RS et al, 2018; Davies MJ et al 2012). The diagnosis, as well as management of complicated facial fractures, is challenging even to the most experienced oral and maxillofacial surgeons, while the presence of coexistent injuries and the complexity of these injuries make it more difficult to consolidate experience and develop realistic treatment protocols. Furthermore, the lack of sufficient specialist facial trauma units results in unacceptable delays from referral to operation, complicating the management and compromising the outcome. Coordination of trauma teams, emergency room physicians, and surgical teams such as neurosurgeons, orthopaedic is vital for the early stabilization and treatment of patients with facial bone fracture (Wong NH et al, 2012; Davies MJ et al, 2012; Follmar KE et al,2007; Van Hout WM et al ,2013, Kostakis G et al, 2012). These injuries may cause serious functional, psychological, physical, and cosmetic disabilities (Kim JW et al 2015; Zachariades N et al 1993) .

The epidemiology of oral and maxillofacial trauma varies from one geographical region to another and even within the same region depending on the many risk factors such as demographic, socioeconomic, cultural, personal behaviour, mental status and environmental factors ( Mathog RH et al, 2000; Fasola AO et al, 2003;Branas CC et al, 2004; Li Z and Li ZB, 2008 ). The common causes worldwide are road traffic accidents (20-83%) (Lee JH et al, 2010; Karagozoglu KH et al, 2012; Walker TW et al 2013; Forouzanfar T et al. 2013; Mijiti A et al, 2014;Jung CP et al, 2016 ); assault( 18- 79%) (Ugboko VI et al 1998; Laskin DM and Best AM, 2000; Olasoji HO et al, 2002; Adebayo ET et al ,2003; Al Ahmed HE et al, 2004; Brasileiro BF et al, 2006; Lee K, 2009a; Lee KH, 2009b; Mijiti A et al, 2014), falls( 10-17% ) (Shankar AN et al, 2012; Van den Bergh B et al 2012; Salentijn EG et al, 2013; Mijiti A et al, 2014), sport injuries (3-7% ) (Bamjee Y et al, 1996; Qudah MA et al, 2002; Al-Khateeb T et al 2007; Bakardjiev A et al, 2007; de Matos FP et al 2010) , hit by moving object ( 5- 15%) (Sakr K, Farag IA et al 2006; Subhashraj K et al, 2007; Thorén H et al, 2010; Chrcanovic BR et al, 2012), bicycle accident ( 2-28% ) (Gomes PP et al, 2006; Kotecha S et al, 2008; Lee JH et al, 2010; Forouzanfar T et al, 2013) , work-related accident (1.7-7% ) (Gassner R et al 2003; Qing-Bin Z et al, 2013) and miscellaneous ( 1.3 %) include pathological fractures, blast injuries, animal attack accident, tooth extraction, and unknown etiology.

Facial bone fractures are a large public health problem with a significant negative impact on an individual's overall health and even survival (Kim JW et al , 2015; Kovacs G, Sowers N, 2018; Prathigudupu RS et al, 2018) . Addressing socio-cultural issues, reviewing and improving road safety legislation, enforcing infrastructure and vehicle standards, and improving post-crash care remain critical to preventing avoidable deaths and disabilities caused by road crashes - which continue to be a major public health challenge ( Mathog RH et al, 2010; Kim JW et al, 2015). Despite the legislative changes and preventative measures involving seatbelt and airbag use, as well as the reduction of drinking and driving, road traffic accidents are still the major cause of facial fractures in many developing countries.

This part of the country ( Provinces 2), is the second most populous province of the country Nepal, located in the central south of the country spans over 9,661 km2 (3,730 sq mi), with a 5,404,145 population of (according to the CBS 2015 year census). Majority of people are poor (48%), illiterates 32% overall and major source of income is agriculture and foreign worker (Wikipedia, 2019). It borders with Bihar states of India. Among the many factors social and cultural similarity, the people of Bihar is presented in this regional hospital for treatment. The road, a major means of transportation here but the condition of the road is very bad.

The main purpose of this study is to investigate the epidemiological characteristics of prevalence, aetiology, sex and age distributions, fracture site, treatment pattern, associated injuries, and complications of maxillofacial fractures treated at the National Medical College and others Hospitals of Birgunj Metropolitan city over a 10-year period from June 2011 to June

Statement of the Problem and Rationale / Justification:

A clearer understanding of the demographic patterns of maxillofacial injuries will assist health care providers as they plan and manage the treatment of traumatic maxillofacial injuries (Al Ahmed et al., 2004; Lee K, 2009; Mijiti A et al., 2014). Such epidemiological information can also be used to guide the future funding of public health programs geared towards prevention.

Understanding maxillofacial trauma helps to evaluate the behaviour patterns of people in different countries and to establish effective prevention and treatment strategies (Maliska et al., 2009; Katarzyna B, Piotr A 2010).

Understanding the cause, severity, and temporal distribution of maxillofacial trauma can assist in establishing clinical and research priorities for effective treatment and prevention of these injuries (Gassner et al., 2003; Qing-Bin Z et al., 2013).

To this end, numerous studies have been carried out to explore the epidemiological features of maxillofacial fractures in different population groups (Ugboko VI et al., 1998; Kieser J et al., 2002; Olasoji HO et al., 2002; Qudah MA et al., 2002; Fasola AO et al., 2003; Al Ahmed HE et al., 2004; Ansari MH., 2004; Gomes PP et al., 2006; Sakr K et al., 2006; Al-Khateeb T et al., 2017; Bakardjiev A et al., 2007; Lee JH et al., 2010; Walker TW et al., 2012; Forouzanfar T et al., 2013; Qing-Bin Z et al., 2013; Van Hout WM et al., 2013; Mijiti A et al., 2014; Jung CP et al., 2016; Nogami S et al., 2019). However, to best our knowledge, there is a lack of reports detailing the causes, incidence, and treatment pattern of maxillofacial injuries, and no study has been published about oral and maxillofacial injuries analysis for this region.

ELIGIBILITY:
Inclusion Criteria:

1. Among the patients have admitted in study sites hospital, those medical records have been maintained (not lost).
2. Patients who had seen by the investigator and had maintained a minimum of 6 weeks of follow-up for retrospective study.

Exclusion Criteria:

1. Patients who had only minor superficial soft tissue injuries which did not require admission.
2. Patients with others fracture only and are not associated with facial injuries like isolated cranial fracture or extremities fracture.
3. Patients with diagnoses different from traumatic fractures, treated by non-surgical means or other surgeons, operated for surgical sterilization purposes or for correction of previous trauma sequelae.
4. Patients whose records were lost, incomplete or illegible.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patients sustain with oral and maxillofacial injuries from the target population brought to study site hospital for advance health care. The patients have been examined, admitted and treated between study duration (10 years) will be enrolled into two-time frames separately. The patient will be identified using the ED case report file (injury report file) or operation registration database.
Sampling Method: Probability Sample
Enrollment: 1030 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Determination of causes and risk factors of oral and maxillofacial injuries | 2019-2021
  This is a pro-retrospective observational study of oral and maxillofacial injuries, is a large public health problem with a significant negative impact on an individual's overall health and even survival. A gender, age, marital status, ethnicity, address, education, occupation, socioeconomically status are variables of trauma. These parameters will be documented in a special form called oral and maxillofacial proforma which is standard, reliable and valid format exceeds the current minimum requirements for clinical governance, addresses and improves the amount of data that is recorded and disseminated during handover.

SECONDARY OUTCOMES:
The role of the health care provider in the management of oral and maxillofacial injuries. | 2019-2021
  Multidisciplinary approaches are required to manage oral and maxillofacial injuries because mainly associated with other injuries. The primary survey is very important to preserve the life of the patients ie ABCDE. Definite management is performed only after proper diagnosis on the basis of clinical or radiological examination, or both. A facial fracture is documented as a standard classification of the zygoma, the accompanying ipsilateral orbital fracture. In the case of a Le Fort II or III fracture, the accompanying nasal and orbital fractures are documented separately.
  Information about the method of treatment will be gathered from the operating notes and will be categorised as open reduction and internal fixation, intermaxillary fixation, reposition without fixation, or orbital floor repair. Other injuries are categorised as neurotrauma, spinal trauma, orthopaedic trauma, general surgical trauma, and other trauma.
Early and late morbidity and mortality assessment in oral and maxillofacial trauma . | 2019-2021
  Early and late complication associated with oral and maxillofacial injury are seen in many circumstances in a period of time. Treatment-Related Adverse Events as Assessed by in trauma. In this study, participants would be followed up 2nd, 6th, 12th, 24th, 48th, 72 and 96th week postoperative. The proforma is used for documentation of complication.

CONTACTS AND LOCATIONS:
Overall Officials: Saroj P Deo, Principal Investigator — National Medical College, Birgunj, Nepal
Locations (1):
- Dr Saroj Prasad Deo, Birgunj, Madhesh, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Data collection to proforma that can be shared with the researcher in the world.
Supporting Information: SAP
Time Frame: As soon I will collect the data of participants of this study, I will upload in the database. then after the completion of this study, it can be shared.
Access Criteria: Only the result of this study.

REFERENCES:
- [Background] Adebayo ET, Ajike OS, Adekeye EO. Analysis of the pattern of maxillofacial fractures in Kaduna, Nigeria. Br J Oral Maxillofac Surg. 2003 Dec;41(6):396-400. doi: 10.1016/s0266-4356(03)00165-7. PMID 14614869
- [Background] Al Ahmed HE, Jaber MA, Abu Fanas SH, Karas M. The pattern of maxillofacial fractures in Sharjah, United Arab Emirates: a review of 230 cases. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Aug;98(2):166-70. doi: 10.1016/j.tripleo.2004.01.020. PMID 15316543
- [Background] Al-Khateeb T, Abdullah FM. Craniomaxillofacial injuries in the United Arab Emirates: a retrospective study. J Oral Maxillofac Surg. 2007 Jun;65(6):1094-101. doi: 10.1016/j.joms.2006.09.013. PMID 17517291
- [Background] Branas CC, Nance ML, Elliott MR, Richmond TS, Schwab CW. Urban-rural shifts in intentional firearm death: different causes, same results. Am J Public Health. 2004 Oct;94(10):1750-5. doi: 10.2105/ajph.94.10.1750. PMID 15451745
- [Background] Bamjee Y, Lownie JF, Cleaton-Jones PE, Lownie MA. Maxillofacial injuries in a group of South Africans under 18 years of age. Br J Oral Maxillofac Surg. 1996 Aug;34(4):298-302. doi: 10.1016/s0266-4356(96)90006-6. PMID 8866064
- [Background] Brasileiro BF, Passeri LA. Epidemiological analysis of maxillofacial fractures in Brazil: a 5-year prospective study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Jul;102(1):28-34. doi: 10.1016/j.tripleo.2005.07.023. Epub 2006 Mar 22. PMID 16831669
- [Background] Boffano P, Roccia F, Gallesio C, Karagozoglu KH, Forouzanfar T. Bicycle-related maxillofacial injuries: a double-center study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Sep;116(3):275-80. doi: 10.1016/j.oooo.2013.03.004. Epub 2013 May 7. PMID 23663988
- [Background] Boffano P, Roccia F, Zavattero E, Dediol E, Uglesic V, Kovacic Z, Vesnaver A, Konstantinovic VS, Petrovic M, Stephens J, Kanzaria A, Bhatti N, Holmes S, Pechalova PF, Bakardjiev AG, Malanchuk VA, Kopchak AV, Galteland P, Mjoen E, Skjelbred P, Koudougou C, Mouallem G, Corre P, Loes S, Lekven N, Laverick S, Gordon P, Tamme T, Akermann S, Karagozoglu KH, Kommers SC, Forouzanfar T. European Maxillofacial Trauma (EURMAT) project: a multicentre and prospective study. J Craniomaxillofac Surg. 2015 Jan;43(1):62-70. doi: 10.1016/j.jcms.2014.10.011. Epub 2014 Oct 22. PMID 25457465
- [Background] Calderoni DR, Guidi Mde C, Kharmandayan P, Nunes PH. Seven-year institutional experience in the surgical treatment of orbito-zygomatic fractures. J Craniomaxillofac Surg. 2011 Dec;39(8):593-9. doi: 10.1016/j.jcms.2010.11.018. Epub 2010 Dec 30. PMID 21195624
- [Background] Chrcanovic BR, Abreu MH, Freire-Maia B, Souza LN. 1,454 mandibular fractures: a 3-year study in a hospital in Belo Horizonte, Brazil. J Craniomaxillofac Surg. 2012 Feb;40(2):116-23. doi: 10.1016/j.jcms.2011.03.012. Epub 2011 Mar 31. PMID 21458284
- [Background] de Matos FP, Arnez MF, Sverzut CE, Trivellato AE. A retrospective study of mandibular fracture in a 40-month period. Int J Oral Maxillofac Surg. 2010 Jan;39(1):10-5. doi: 10.1016/j.ijom.2009.10.005. Epub 2009 Nov 14. PMID 19914802
- [Background] Davies MJ, Wells C, Squires PA, Hodgetts TJ, Lecky FE. Civilian firearm injury and death in England and Wales. Emerg Med J. 2012 Jan;29(1):10-4. doi: 10.1136/emj.2009.085837. Epub 2011 Nov 4. PMID 22058090
- [Background] Fasola AO, Nyako EA, Obiechina AE, Arotiba JT. Trends in the characteristics of maxillofacial fractures in Nigeria. J Oral Maxillofac Surg. 2003 Oct;61(10):1140-3. doi: 10.1016/s0278-2391(03)00671-2. PMID 14586847
- [Background] Follmar KE, Debruijn M, Baccarani A, Bruno AD, Mukundan S, Erdmann D, Marcus JR. Concomitant injuries in patients with panfacial fractures. J Trauma. 2007 Oct;63(4):831-5. doi: 10.1097/TA.0b013e3181492f41. PMID 18090013
- [Background] Forouzanfar T, Salentijn E, Peng G, van den Bergh B. A 10-year analysis of the "Amsterdam" protocol in the treatment of zygomatic complex fractures. J Craniomaxillofac Surg. 2013 Oct;41(7):616-22. doi: 10.1016/j.jcms.2012.12.004. Epub 2013 Jan 30. PMID 23375533
- [Background] Gassner R, Tuli T, Hachl O, Rudisch A, Ulmer H. Cranio-maxillofacial trauma: a 10 year review of 9,543 cases with 21,067 injuries. J Craniomaxillofac Surg. 2003 Feb;31(1):51-61. doi: 10.1016/s1010-5182(02)00168-3. PMID 12553928
- [Background] Gomes PP, Passeri LA, Barbosa JR. A 5-year retrospective study of zygomatico-orbital complex and zygomatic arch fractures in Sao Paulo State, Brazil. J Oral Maxillofac Surg. 2006 Jan;64(1):63-7. doi: 10.1016/j.joms.2005.09.012. PMID 16360858
- [Background] Imholz B, Combescure C, Scolozzi P. Is age of the patient an independent predictor influencing the management of cranio-maxillo-facial trauma? A retrospective study of 308 patients. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Jun;117(6):690-6. doi: 10.1016/j.oooo.2014.03.010. Epub 2014 Mar 24. PMID 24842446
- [Background] Johnson J, Markiewicz MR, Bell RB, Potter BE, Dierks EJ. Gun orientation in self-inflicted craniomaxillofacial gunshot wounds: risk factors associated with fatality. Int J Oral Maxillofac Surg. 2012 Aug;41(8):895-901. doi: 10.1016/j.ijom.2012.05.013. Epub 2012 Jun 20. PMID 22727362
- [Background] Jung CP, Tsai AI, Chen CM. A 2-year retrospective study of pediatric dental emergency visits at a hospital emergency center in Taiwan. Biomed J. 2016 Jun;39(3):207-13. doi: 10.1016/j.bj.2016.06.004. Epub 2016 Aug 9. PMID 27621123
- [Background] Kieser J, Stephenson S, Liston PN, Tong DC, Langley JD. Serious facial fractures in New Zealand from 1979 to 1998. Int J Oral Maxillofac Surg. 2002 Apr;31(2):206-9. doi: 10.1054/ijom.2002.0208. PMID 12102421
- [Background] Kotecha S, Scannell J, Monaghan A, Williams RW. A four year retrospective study of 1,062 patients presenting with maxillofacial emergencies at a specialist paediatric hospital. Br J Oral Maxillofac Surg. 2008 Jun;46(4):293-6. doi: 10.1016/j.bjoms.2007.11.011. Epub 2008 Jan 4. PMID 18177983
- [Background] Bogusiak K, Arkuszewski P. Characteristics and epidemiology of zygomaticomaxillary complex fractures. J Craniofac Surg. 2010 Jul;21(4):1018-23. doi: 10.1097/scs.0b013e3181e62e47. PMID 20677370
- [Background] van den Bergh B, Karagozoglu KH, Heymans MW, Forouzanfar T. Aetiology and incidence of maxillofacial trauma in Amsterdam: a retrospective analysis of 579 patients. J Craniomaxillofac Surg. 2012 Sep;40(6):e165-9. doi: 10.1016/j.jcms.2011.08.006. Epub 2011 Sep 14. PMID 21917471
- [Background] Kostakis G, Stathopoulos P, Dais P, Gkinis G, Igoumenakis D, Mezitis M, Rallis G. An epidemiologic analysis of 1,142 maxillofacial fractures and concomitant injuries. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Nov;114(5 Suppl):S69-73. doi: 10.1016/j.tripleo.2011.08.029. Epub 2012 Feb 28. PMID 23083959
- [Background] Kim JW, Wu J, Shen SG, Xu B, Shi J, Zhang S. Interdisciplinary Surgical Management of Multiple Facial Fractures With Image-Guided Navigation. J Oral Maxillofac Surg. 2015 Sep;73(9):1767-77. doi: 10.1016/j.joms.2015.03.029. Epub 2015 Mar 20. PMID 25869985
- [Background] Laskin DM, Best AM. Current trends in the treatment of maxillofacial injuries in the United States. J Oral Maxillofac Surg. 2000 Feb;58(2):207-15. doi: 10.1016/s0278-2391(00)90341-0. PMID 10670601
- [Background] Li Z, Li ZB. Characteristic changes of pediatric maxillofacial fractures in China during the past 20 years. J Oral Maxillofac Surg. 2008 Nov;66(11):2239-42. doi: 10.1016/j.joms.2007.12.032. PMID 18940486
- [Background] Lee K. Trend of alcohol involvement in maxillofacial trauma. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Apr;107(4):e9-13. doi: 10.1016/j.tripleo.2008.12.020. Epub 2009 Feb 8. PMID 19201626
- [Background] Lee KH. Interpersonal violence and facial fractures. J Oral Maxillofac Surg. 2009 Sep;67(9):1878-83. doi: 10.1016/j.joms.2009.04.117. PMID 19686924
- [Background] Lee JH, Cho BK, Park WJ. A 4-year retrospective study of facial fractures on Jeju, Korea. J Craniomaxillofac Surg. 2010 Apr;38(3):192-6. doi: 10.1016/j.jcms.2009.06.002. Epub 2009 Jul 3. PMID 19577480
- [Background] Mijiti A, Ling W, Tuerdi M, Maimaiti A, Tuerxun J, Tao YZ, Saimaiti A, Moming A. Epidemiological analysis of maxillofacial fractures treated at a university hospital, Xinjiang, China: A 5-year retrospective study. J Craniomaxillofac Surg. 2014 Apr;42(3):227-33. doi: 10.1016/j.jcms.2013.05.005. Epub 2013 Jun 19. PMID 23791439
- [Background] Mathog RH, Toma V, Clayman L, Wolf S. Nonunion of the mandible: an analysis of contributing factors. J Oral Maxillofac Surg. 2000 Jul;58(7):746-52; discussion 752-3. doi: 10.1053/joms.2000.7258. PMID 10883689
- [Background] Nogami S, Yamauchi K, Bottini GB, Otake Y, Sai Y, Morishima H, Higuchi K, Ito K, Gaggl A, Takahashi T. Fall-related mandible fractures in a Japanese population: A retrospective study. Dent Traumatol. 2019 Jun;35(3):194-198. doi: 10.1111/edt.12471. Epub 2019 Apr 29. PMID 30916458
- [Background] Olasoji HO, Tahir A, Arotiba GT. Changing picture of facial fractures in northern Nigeria. Br J Oral Maxillofac Surg. 2002 Apr;40(2):140-3. doi: 10.1054/bjom.2001.0716. PMID 12180207
- [Background] Jose A, Nagori SA, Agarwal B, Bhutia O, Roychoudhury A. Management of maxillofacial trauma in emergency: An update of challenges and controversies. J Emerg Trauma Shock. 2016 Apr-Jun;9(2):73-80. doi: 10.4103/0974-2700.179456. PMID 27162439
- [Background] Qudah MA, Bataineh AB. A retrospective study of selected oral and maxillofacial fractures in a group of Jordanian children. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2002 Sep;94(3):310-4. doi: 10.1067/moe.2002.127406. PMID 12324784
- [Background] Qing-Bin Z, Zhao-Qiang Z, Dan C, Yan Z. Epidemiology of maxillofacial injury in children under 15 years of age in southern China. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Apr;115(4):436-41. doi: 10.1016/j.oooo.2012.04.026. Epub 2012 Aug 31. PMID 22940023
- [Background] Roccia F, Savoini M, Ramieri G, Zavattero E. An analysis of 711 victims of interpersonal violence to the face, Turin, Italy. J Craniomaxillofac Surg. 2016 Aug;44(8):1025-8. doi: 10.1016/j.jcms.2016.05.021. Epub 2016 Jun 6. PMID 27328893
- [Background] Sakr K, Farag IA, Zeitoun IM. Review of 509 mandibular fractures treated at the University Hospital, Alexandria, Egypt. Br J Oral Maxillofac Surg. 2006 Apr;44(2):107-11. doi: 10.1016/j.bjoms.2005.03.014. PMID 15896887
- [Background] Subhashraj K, Nandakumar N, Ravindran C. Review of maxillofacial injuries in Chennai, India: a study of 2748 cases. Br J Oral Maxillofac Surg. 2007 Dec;45(8):637-9. doi: 10.1016/j.bjoms.2007.03.012. Epub 2007 May 23. PMID 17524534
- [Background] Salentijn EG, van den Bergh B, Forouzanfar T. A ten-year analysis of midfacial fractures. J Craniomaxillofac Surg. 2013 Oct;41(7):630-6. doi: 10.1016/j.jcms.2012.11.043. Epub 2013 Feb 15. PMID 23419413
- [Background] Thoren H, Snall J, Salo J, Suominen-Taipale L, Kormi E, Lindqvist C, Tornwall J. Occurrence and types of associated injuries in patients with fractures of the facial bones. J Oral Maxillofac Surg. 2010 Apr;68(4):805-10. doi: 10.1016/j.joms.2009.09.057. Epub 2010 Jan 15. PMID 20079962
- [Background] Tuli T, Haechl O, Berger N, Laimer K, Jank S, Kloss F, Brandstatter A, Gassner R. Facial trauma: how dangerous are skiing and snowboarding? J Oral Maxillofac Surg. 2010 Feb;68(2):293-9. doi: 10.1016/j.joms.2009.09.072. PMID 20116698
- [Background] van Hout WM, Van Cann EM, Abbink JH, Koole R. An epidemiological study of maxillofacial fractures requiring surgical treatment at a tertiary trauma centre between 2005 and 2010. Br J Oral Maxillofac Surg. 2013 Jul;51(5):416-20. doi: 10.1016/j.bjoms.2012.11.002. Epub 2012 Dec 4. PMID 23218202
- [Background] Walker TW, Byrne S, Donnellan J, McArdle N, Kerin MJ, McCann PJ. West of Ireland facial injury study. Part 1. Br J Oral Maxillofac Surg. 2012 Oct;50(7):631-5. doi: 10.1016/j.bjoms.2011.09.025. Epub 2011 Dec 20. PMID 22192609
- [Background] Walker TW, Donnellan J, Byrne S, McArdle N, Kerin MJ, McCann PJ. West of Ireland facial injury study. Part 2. Br J Oral Maxillofac Surg. 2012 Oct;50(7):e99-e103. doi: 10.1016/j.bjoms.2011.09.026. Epub 2012 Mar 17. PMID 22425017
- [Background] Yamamoto K, Matsusue Y, Horita S, Murakami K, Sugiura T, Kirita T. Maxillofacial fractures sustained in bicycle accidents. J Oral Maxillofac Surg. 2011 Jun;69(6):e155-60. doi: 10.1016/j.joms.2010.12.028. Epub 2011 Apr 15. PMID 21496994
- [Background] Zachariades N, Papademetriou I, Rallis G. Complications associated with rigid internal fixation of facial bone fractures. J Oral Maxillofac Surg. 1993 Mar;51(3):275-8; discussion 278-9. doi: 10.1016/s0278-2391(10)80174-0. PMID 8445470
- See also: The top 10 causes of death; fact-sheets. — https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death